CLINICAL TRIAL: NCT00005868
Title: Taxotere and Cisplatin as Induction Chemotherapy in Patients With Stage IIIa N2 Non Small Cell Lung Cancer (NSCLC)
Brief Title: Docetaxel and Cisplatin in Treating Patients With Untreated Stage IIIA Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-08984; EORTC-08984
Record Dates: First submitted 2000-06-02; First posted 2003-05-21 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of docetaxel and cisplatin in treating patients who have untreated stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the therapeutic activity of docetaxel and cisplatin in patients with untreated stage IIIA non-small cell lung cancer.
* Determine the safety of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour on day 1 and cisplatin IV over 30 minutes on days 1 and 2. Treatment continues every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 24-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IIIA non-small cell lung cancer (NSCLC) (T1-3, N2, M0)

  * Unresectable metastasis to ipsilateral mediastinal and/or subcarinal lymph nodes
* Measurable disease

  * Must be at least 20 mm in one dimension by conventional techniques or at least 10 mm by spiral CT scan
* No distant metastases
* No CNS involvement
* No pleural or pericardial effusion

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* AST/ALT no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.25 ULN
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No superior vena cava syndrome
* No uncontrolled congestive heart failure or angina
* No myocardial infarction within past year
* No uncontrolled hypertension or arrhythmia

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent active infection requiring IV antibiotic therapy
* No other prior malignancy in past 5 years except carcinoma in situ of the cervix or adequately treated basal cell carcinoma, excluding melanoma, breast cancer, and hypernephroma
* No concurrent illness or medical condition which is a contraindication for corticosteroid therapy (e.g., active ulcer, unstable diabetes mellitus)
* No motor or sensory neurotoxicity of grade 2 or greater
* No psychological, familial, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* No prior chemotherapy for NSCLC
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy

Radiotherapy:

* No prior radiotherapy for NSCLC
* No concurrent radiotherapy

Surgery:

* No prior surgery for NSCLC

Other:

* At least 1 month since prior investigational agents
* No other concurrent experimental medications

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2000-03; Primary Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, MD, PhD, Study Chair — Free University Medical Center
Locations (23):
- Thoraxklinik Rohrbach, Heidelberg, Germany
- Italy (2):
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova)
  - Oncologia Medica - Perugia, Perugia
- Netherlands (17):
  - Leyenburg Ziekenhuis, 's-Gravenhage (Den Haag, the Hague)
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Slotervaart Ziekenhuis, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Longarts Dr. J.M. Smit Rynstate Hospital, Arnhem
  - Ziekenhuis St Jansdal, Harderwijk
  - Leiden University Medical Center, Leiden
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - University Medical Center Nijmegen, Nijmegen
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Twee Steden Ziekenhuis Vestiging Tilburg, Tilburg
  - Academisch Ziekenhuis Utrecht, Utrecht
  - Zaas Medisch Centrum, Zaandam
  - Sophia Ziekehuis, Zwolle
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- United Kingdom (2):
  - Weston Park Hospital, Sheffield, England
  - Royal Marsden Hospital, Sutton, England

REFERENCES:
- [Result] Biesma B, Manegold C, Smit HJ, Willems L, Legrand C, Passioukov A, van Meerbeeck JP, Giaccone G; EORTC Lung Cancer Group. Docetaxel and cisplatin as induction chemotherapy in patients with pathologically-proven stage IIIA N2 non-small cell lung cancer: a phase II study of the European organization for research and treatment of cancer (EORTC 08984). Eur J Cancer. 2006 Jul;42(10):1399-406. doi: 10.1016/j.ejca.2006.01.049. Epub 2006 Jun 8. PMID 16759850
- [Result] Manegold C, Biesma B, Smit H, et al.: Docetaxel and cisplatin as induction chemotherapy in stage IIIA N2 non-small cell lung cancer (NSCLC): an EORTC phase II trial (08984). [Abstract] J Clin Oncol 22 (Suppl 14): A-7166, 657s, 2004.
- [Result] Manegold C, Biesma B, Debruyne C, et al.: Docetaxel and cisplatin as induction chemotherapy in stage IIIA N2 non-small cell lung cancer (NSCLC): an EORTC phase II trial (08984). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-2719, 2002.